CLINICAL TRIAL: NCT00635258
Title: Administration of GnRH Antagonist to Oocyte Donation Recipients During Endometrial Preparation.
Brief Title: Administration of GnRH Antagonist to Oocyte Donation Recipients
Acronym: GnRH-Ovodon
Status: Completed | Type: Observational
Sponsor: Centro Ginecologia y Obstetricia. (Other)
Collaborators: University of Valencia (Other)
Responsible Party: Fernando Bonilla-Musoles, CEGIOB
Other Study IDs: GnRH-ant.Ovodon
Record Dates: First submitted 2008-02-26; First posted 2008-03-13 (Estimated); Last update posted 2008-03-13 (Estimated); Status verified 2008-03

CONDITIONS: Pregnancy; Embryo Implantation
Keywords: GnRH antagonist; oocyte donation; pregnancy; implantation
MeSH Terms: interventions — Triptorelin Pamoate; Gonadotropin-Releasing Hormone; ganirelix; LHRH, Ac-Nal(1)-Cpa(2)-Trp(3)-Arg(6)-Ala(10)-

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- GnRH-ant: Patients were treated with a GnRH antagonist (Orgalutran®; 0,25 mg/d, sc.) commencing on day 1 of the menstrual cycle and maintained until the day of donor's hCG administration.
  Interventions: Drug: GnRH antagonist (Orgalutran®)
- GnRH-a: GnRH long protocol using 0.1 mg/day triptorelin s.c (Decapeptyl®, Ipsen Pharma, Barcelona, Spain) was started on day 21-24 of the preceding cycle for at least 14 days to produce an agonadal state. Furthermore, the triptorelin administration was maintained until the day of donor's hCG administration.
  Interventions: Drug: triptorelin (Decapeptyl®, Ipsen Pharma, Barcelona, Spain)

INTERVENTIONS:
Drug: triptorelin (Decapeptyl®, Ipsen Pharma, Barcelona, Spain) — 0.1 mg/day triptorelin s.c (Decapeptyl®, Ipsen Pharma, Barcelona, Spain) was started on day 21-24 of the preceding cycle for at least 14 days to produce an agonadal state.
  Other Names: GnRH agonist
  Groups: GnRH-a
Drug: GnRH antagonist (Orgalutran®) — GnRH antagonist (Orgalutran®; 0,25 mg/d, sc.) commencing on day 1 of the menstrual cycle and maintained until the day of donor's hCG administration.
  Other Names: GnRH antagonist
  Groups: GnRH-ant

SUMMARY:
This prospective and randomized study was performed to evaluate whether the replacement of GnRH agonist by a GnRH antagonist in oocyte donation recipients during endometrial preparation has any impact on pregnancy and implantation rates.

DETAILED DESCRIPTION:
This was a prospective and randomized study undertaken between January 2004 and December 2007. One hundred patients with an indication for oocyte donation with functioning ovaries and IVF with or without intracytoplasmatic sperm injection (ICSI) were recruited for the study. After assignment to IVF or IVF/ICSI randomization was performed to 1 of the 2 treatment groups (GnRH agonist or GnRH antagonist during endometrial preparation in oocyte donation recipients) using a computed-generated randomization schedule assigned via numbered sealed envelopes.

In our program, we used excess oocytes from IVF that were voluntarily donated by patients after informed consent.

The indications for oocyte donation were reduced ovarian reserve (59%), recurrent IVF failures (21%), premature ovarian failure (16%), and genetic anomaly (4%).

This study was performed according to the declaration of Helsinki and the European Community note on Good Clinical Practice for trials on medical products in the European Community (CPMP Working Party on Efficacy of Medical Products, 1990). Furthermore, the local ethics committee approved the study protocol, and written informed consent was obtained from all patients.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18-34 years
* Body mass index between 19-30 kg/m2;
* History of regular menstrual cycles, ranging from 25-35 days
* No relevant systemic disease (all patients were screened for hepatitis B and C, human immunodeficiency viruses I and II, syphylis, and vaginal infection), genetic disease, severe endometriosis or pelvic inflamatory disease
* No more than two previous IVF cycles; and
* No previous IVF cycles with poor response (less than three oocytes in a previous IVF cycle) or severe ovarian hyperstimulation syndrome.

Exclusion Criteria:

* Patients without inclusion criteria.

Ages: 18 Years to 34 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Patients with an indication for oocyte donation with functioning ovaries.
Sampling Method: Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2004-01; Primary Completion 2007-12 (Actual); Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
pregnancy and implantation rates | "at 7 weeks"

SECONDARY OUTCOMES:
age of the recipients, body mass index, days undergoing oestrogen therapy | "at 1 mounth"

CONTACTS AND LOCATIONS:
Overall Officials: Raga Francisco, M.D., Ph.D., Principal Investigator — Centro Ginecologia y Obstetricia.
Locations (1):
- CEGIOB, Valencia, Valencia, Spain

REFERENCES:
- [Background] Casan EM, Raga F, Bonilla-Musoles F, Polan ML. Human oviductal gonadotropin-releasing hormone: possible implications in fertilization, early embryonic development, and implantation. J Clin Endocrinol Metab. 2000 Apr;85(4):1377-81. doi: 10.1210/jcem.85.4.6503. PMID 10770169
- [Background] Raga F, Casan EM, Kruessel J, Wen Y, Bonilla-Musoles F, Polan ML. The role of gonadotropin-releasing hormone in murine preimplantation embryonic development. Endocrinology. 1999 Aug;140(8):3705-12. doi: 10.1210/endo.140.8.6899. PMID 10433230
- [Background] Casan EM, Raga F, Polan ML. GnRH mRNA and protein expression in human preimplantation embryos. Mol Hum Reprod. 1999 Mar;5(3):234-9. doi: 10.1093/molehr/5.3.234. PMID 10333357
- [Background] Raga F, Casan EM, Wen Y, Huang HY, Bonilla-Musoles F, Polan ML. Independent regulation of matrix metalloproteinase-9, tissue inhibitor of metalloproteinase-1 (TIMP-1), and TIMP-3 in human endometrial stromal cells by gonadotropin-releasing hormone: implications in early human implantation. J Clin Endocrinol Metab. 1999 Feb;84(2):636-42. doi: 10.1210/jcem.84.2.5464. PMID 10022430
- [Background] Raga F, Casan EM, Kruessel JS, Wen Y, Huang HY, Nezhat C, Polan ML. Quantitative gonadotropin-releasing hormone gene expression and immunohistochemical localization in human endometrium throughout the menstrual cycle. Biol Reprod. 1998 Sep;59(3):661-9. doi: 10.1095/biolreprod59.3.661. PMID 9716567